CLINICAL TRIAL: NCT06318507
Title: The Intestinal Microbiome in Triple Negative Breast Cancer Treated with Immunotherapy
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Justin Brown, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-014
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: Fecal microbial diversity — Fecal microbiome diversity via 16S rRNA and metagenomic sequencing

SUMMARY:
This study will determine how the intestinal microbiome differs between patients with obesity and early triple-negative breast cancer who achieve a pathologic complete response from preoperative anti-PD-1 immunotherapy (pembrolizumab) versus patients who do not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Female biological sex
* Newly diagnosed, previously untreated, histologically confirmed early triple-negative breast cancer
* Plan to initiate preoperative anti-PD-1 immunotherapy using pembrolizumab
* Overweight or obesity, defined as a body mass index >=25 kg/m2
* Ability to provide written informed consent
* Allow the collection and storage of biospecimens and data for future use

Exclusion Criteria:

* Active autoimmune disease
* Concomitant conditions that require the use of antibiotics (e.g., chronic sinusitis)
* Digestive disease disorders (e.g., irritable bowel syndrome, Crohn's disease)
* Currently pregnant, breastfeeding, or planning to become pregnant within the next 24 weeks
* Recent (within 90 days) use of glucocorticoids for more than 10 consecutive days
* Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric, or other condition that, in the investigator's opinion, would preclude participation or successful compliance with the protocol
* Any other situation that, in the opinion of the investigator, would negatively impact subject safety or successful compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of survivors of early triple-negative breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | Week 24
  Defined as ypT0/Tis ypN0, ypT0 ypN0, and ypT0/Tis

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No